CLINICAL TRIAL: NCT04996511
Title: Day Case Colectomy: Optimizing Short Stay-surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Q021
Record Dates: First submitted 2021-05-05; First posted 2021-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal Surgery Patients (Experimental)
  Interventions: Device: PulseOn

INTERVENTIONS:
Device: PulseOn — Postoperative HRV measurement
  Other Names: Faros; Emfit QS

SUMMARY:
HRV measurement of patients recovering from laparoscopic colorectal resection for any pathology.

DETAILED DESCRIPTION:
Patients scheduled for colorectal surgery are recruited to the study. HRV parameters including e.g. RMSSD are evaluated before and after surgery. The effect of surgery and possible complications associated with it on parameters and relationship with specific adverse effects caused by complications are evaluated.

ELIGIBILITY:
Inclusion Criteria:

• Colorectal resection for any pathology

Exclusion Criteria:

• Arrhytmias likely to cause problems with HRV measurements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) change | 3 days
  Reliability of HRV parameters

CONTACTS AND LOCATIONS:
Overall Officials: Juha KA Rinne, MD, Principal Investigator — Päijät Häme Central Hospital
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Finland

REFERENCES:
- [Derived] Rinne JKA, Miri S, Oksala N, Vehkaoja A, Kossi J. Evaluation of a wrist-worn photoplethysmography monitor for heart rate variability estimation in patients recovering from laparoscopic colon resection. J Clin Monit Comput. 2023 Feb;37(1):45-53. doi: 10.1007/s10877-022-00854-w. Epub 2022 Apr 8. PMID 35394583